CLINICAL TRIAL: NCT07244679
Title: The Effect of Sacroiliac Joint Manipulation on Core Stabilization in Healthy Individuals
Brief Title: Sacroiliac Manipulation and Core Stability in Healthy Adults
Acronym: SIJCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Esra BECENI, Lecturer, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BAU-FTR-SIJCORE-2022
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Health Adults; Core Stabilization
Keywords: Sacroiliac Joint Manipulation; Core Stabilization; Chriopractic

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, single-blind, prospective study
Who Masked: Outcomes Assessor
Masking Description: Randomization will be done by sealed envelope method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIJ Manipulation Group (Experimental): Bilateral HVLA SIJ manipulation applied at PSIS
  Interventions: Other: Sacroiliac Joint Manipulation (HVLA)
- Control Group (No Treatment) (No Intervention): Participants received no manipulation; only baseline and post-test evaluations were performed.

INTERVENTIONS:
Other: Sacroiliac Joint Manipulation (HVLA) — HVLA manipulation applied bilaterally at the sacroiliac joint (PSIS) to improve lumbopelvic stability.
  Other Names: Experimental Group
  Arms: SIJ Manipulation Group

SUMMARY:
Sacroiliac joint (SIJ) dysfunction is a common cause of lumbopelvic instability, often linked to altered load transfer between the spine and lower limbs. Although various therapeutic interventions are used to restore joint alignment and improve neuromuscular control, the immediate effects of chiropractic manipulation on core stabilization in asymptomatic individuals remain unclear. This randomized controlled study aimed to examine the acute impact of bilateral sacroiliac joint high-velocity, low-amplitude (HVLA) manipulation on trunk stability in healthy adults. Sixty participants aged 18-40 years were randomly assigned to either a manipulation group or a control group. Core stabilization performance and postural control were evaluated using standardized tests including the Centaur Trunk Training (CTT) biofeedback system, plank, sit-ups endurance, and flexibility assessments. The findings demonstrated significant short-term improvements in trunk stability and flexibility following manipulation, suggesting that sacroiliac joint adjustments may positively influence neuromuscular activation and motor control in healthy individuals.

DETAILED DESCRIPTION:
SIJ is recognized as a key anatomical structure responsible for transmitting mechanical loads between the spine and the lower extremities. Even minor restrictions in SIJ mobility have the potential to alter lumbopelvic alignment, modify core muscle activation patterns, and influence postural stability. Although these alterations may occur in symptomatic and asymptomatic populations alike, the precise neuromuscular mechanisms through which SIJ mobility affects trunk control remain an area of ongoing scientific inquiry.

Manual therapy techniques-particularly HVLA manipulation-are frequently employed to restore joint mobility, regulate proprioceptive input, and optimize neuromuscular coordination within the lumbopelvic region. HVLA manipulation has been proposed to facilitate rapid mechanical and neurophysiological responses, including improved segmental motion, enhanced afferent feedback, and short-term modifications in motor unit recruitment. Despite these proposed mechanisms, empirical evidence concerning the acute effects of SIJ-directed HVLA manipulation in healthy adults is limited.

Core stabilization constitutes another critical component of lumbopelvic rehabilitation. This approach emphasizes the activation, endurance, and coordinated function of deep trunk musculature-particularly the transversus abdominis, multifidus, and associated stabilizer groups-which collectively contribute to spinal alignment and postural equilibrium. Core stabilization strategies are widely supported in theory; however, their interaction with manual therapy techniques, especially in terms of immediate biomechanical and neuromuscular responses, has not been thoroughly examined in healthy individuals.

This randomized controlled trial was designed to investigate the immediate effects of bilateral SIJ HVLA manipulation on trunk stability and postural control in healthy adults. The study was conducted at Ataşehir Florence Nightingale Hospital and included participants aged 18-40 years who met predefined eligibility criteria. After completing baseline assessments, participants were randomly assigned to one of two groups:(1) the SIJ Manipulation Group, which received bilateral HVLA manipulation at the posterior superior iliac spines (PSIS) in a side-lying position, and (2) the Control Group (No Treatment), which completed the same assessment procedures without receiving any therapeutic intervention.

A comprehensive set of outcome measures was selected to evaluate multiple dimensions of lumbopelvic function. Pelvic alignment patterns were examined using the Derifield-Thompson leg check, while lumbar spine mobility was assessed with the Modified Schober Test. Core endurance and trunk muscle performance were measured using standardized sit-up and plank tests. The most detailed assessment was performed with the CTT biofeedback system, an objective device capable of analyzing postural control across 22 angular positions ranging from 0° to ±180°, thereby providing multidimensional insight into trunk stability.

The HVLA manipulation procedure involved a brief, controlled thrust delivered bilaterally to the SIJ region following established clinical guidelines. All post-intervention assessments were performed immediately after the procedure according to the predefined protocol. Ethical approval for the study was obtained from the Istanbul Yeni Yüzyıl University Clinical Research Ethics Committee (Decision No: 24.03.2022/14), and written informed consent was obtained from all participants prior to enrollment.

This trial was designed to explore the theoretical mechanisms through which SIJ manipulation may influence trunk stability, neuromuscular activation, and early postural adjustments in asymptomatic individuals. The findings and statistical outcomes of the study will be reported separately in the Results section of this clinical trial record. The present protocol description is intended solely to outline the scientific rationale, methodological framework, and procedural details of the study, without including any data-driven conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged between 18 and 40 years
* No history of low back or pelvic pain within the last 6 months
* No previous spinal or sacroiliac joint surgery
* No current neurological or musculoskeletal disorders
* Able to maintain standing and sitting positions without discomfort
* Voluntary participation with informed consent

Exclusion Criteria:

* History of chronic low back pain or sacroiliac dysfunction
* Previous fractures, dislocations, or surgery in the lumbopelvic region
* Neurological, vestibular, or systemic disorders affecting balance or movement
* Pregnancy or suspected pregnancy
* Use of pain medication, muscle relaxants, or anti-inflammatory drugs within the last 48 hours
* Contraindications to manual therapy (osteoporosis, malignancy, inflammatory joint disease, acute disc herniation, cauda equina syndrome)
* Refusal or inability to participate in the study protocol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Trunk Stability Index CTT biofeedback system | Baseline (pre-intervention) and immediately after intervention (within 1 week)
  Measurement of trunk stability using the CTT biofeedback system, which evaluates angular deviation and postural control across 22 tilt positions (0° to ±180°). Lower deviation values indicate greater stability.

SECONDARY OUTCOMES:
Static Core Endurance (Plank Test Duration) | Baseline and immediately post-intervention (within 1 week)
  Duration (in seconds) that participants can maintain a standard plank position to assess static trunk endurance. Higher values indicate greater core stability and muscular endurance.
Sit-ups Endurance Test | Baseline and 1 week post-intervention
  Number of sit-ups completed in 60 seconds to evaluate abdominal and hip flexor endurance. Increased repetitions indicate improved muscular performance.
Modified Schober Test (Lumbar Flexibility) | Baseline and post-intervention (1 week)
  Measurement of lumbar spine flexibility in centimeters. The difference between baseline and post-test scores reflects improvement in spinal mobility.
Finger-to-Floor Distance (Trunk Flexibility) | Baseline and post-intervention (1 week)
  Distance (cm) between fingertips and floor during maximal forward flexion. Shorter distance indicates improved flexibility and spinal mobility.
Derifield-Thompson Leg Check Test (Pelvic Alignment) | Baseline and immediately post-intervention
  Manual assessment used to detect leg length discrepancy associated with sacroiliac joint dysfunction. Improvement is noted as reduction in asymmetry between pre- and post-intervention.
Lumbar and Hip Range of Motion (Goniometric Assessment) | Baseline and post-intervention (1 week)
  Active and passive range of motion (degrees) of the lumbar spine and hip joints, measured using a goniometer. Parameters include lumbar flexion, extension, and hip flexion. Greater values indicate increased joint mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataşehir Florence Nightingale Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study was completed as an academic clinical trial involving healthy volunteers. Individual participant data (IPD) will not be shared publicly because the dataset contains identifiable information collected under institutional ethics approval and informed consent restricted to internal analysis. Only aggregate (group-level) results will be available upon publication.